CLINICAL TRIAL: NCT05160337
Title: Clinical Study on Healthy Volunteers for Validating the Stability of Different Diagnostic Biomarkers Studied at Firalis
Brief Title: Validation of the Stability of Diagnostic Biomarkers on Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firalis SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A00405-36
Record Dates: First submitted 2021-11-08; First posted 2021-12-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: biomarkers; chronobiology; healthy volounteers; diagnostic biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volunteers (Other): Healthy Volunteers will be recruited into the study
  Interventions: Diagnostic Test: Biomarker based IVD tests

INTERVENTIONS:
Diagnostic Test: Biomarker based IVD tests — Biomarker based IVD tests

SUMMARY:
Stability studies on the peripheral biomarkers (lncRNAs, sncRNAs, mRNAs, proteins, lipids/metabolites) measured by Firalis IVD test candidates and effect of gender, age, nutrition on their expression level

DETAILED DESCRIPTION:
Firalis SA and its affiliate Amoneta Diagnostics SAS are developing novel in-vitro diagnostic (IVD) tests for diverse diagnostic applications for major human diseases, including cardiovascular, and neurodegenerative disorders. These tests measure in blood and other peripheral body fluids; long non-coding RNAs (lncRNAs), small non-coding RNAs (sncRNAs), messenger RNAs (mRNAs), circulating proteins, lipids and metabolites. In addition, since 2020, Firalis is producing the salivary test EasyCOV for detection of Covid-19 positivity in both symptomatic and asymptomatic subjects. Firalis group is the sponsor of a pipeline of various clinical studies conducted in diverse National and European clinical sites of excellence, enrolling patients affected by the targeted diseases studied such as acute myocardial injury, Alzheimer disease for the proof of performance phase of the biomarkers and IVD test candidates. The present specific study aims to collect biological samples to complete the analytical validation of its diverse IVD tools namely the evaluation of the stability of the biomarkers and the effect of age, gender, nutrition and inter-period on the expression level of the studied biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Participants who sign the informed consent forms for sample collection and data collection both anonymized and reported in CRF.
* Able to comply with all study procedures.
* Healthy Volunteers having no apparent disease.
* Adults, both genders, aged 18-85 years.
* Participants with no apparent motor or mental health abnormality.
* Participants having no major disabling mental or physical disability that would require hospitalization.
* Body weight above 50 kg if male, above 40 kg if female.

Exclusion Criteria:

* Any subject who did not sign the Informed Consent form.
* Any subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any subject in the exclusion period of a previous study according to applicable regulations.
* Any subject who cannot be contacted in case of emergency.
* Any subject who is the Investigator or any sub-investigator, research assistant, study coordinator, or other staff thereof, directly involved in the conduct of the protocol.
* Any subject with a disease that, in the judgement of the investigator, would interfere with the conduct of study or harm the safety of volunteer.
* Subjects with disabling disease or abnormal health status are excluded.
* Subjects aged below 18 years and older than 85 years are excluded.
* Pregnant, parturient and nursing women are excluded.
* Subjects deprived of their liberty by a judicial or administrative decision, protected adults and vulnerable persons are excluded.
* Subjects who are under legal protection or who are unable to express their consent are not included.
* Any subject who reports in the questionnaire of the screening period having one of the following diseases is excluded:

  * Any psychiatric or neurodegenerative disease or neurologic disorder.
  * Hypertension.
  * Any cardiovascular disease.
  * Any chronic inflammatory disease such as rheumatoid arthritis.
  * Any cancer.
  * Frequent headaches and/or migraine, recurrent nausea and/or vomiting.
* Any subject who did a blood donation, any volume, within 2 months before inclusion.
* Any subject who reports in the questionnaire of the screening period having medication(s) for one or more of the above diseases is excluded.
* Drug or alcohol abuse or smoking more than 10 cigarettes or equivalent.
* Subjects with no apparent disease and symptoms, but with unknown Covid-19 positivity are not excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
lncRNA Biomarker expression before breakfast intake | T0- Baseline in the morning before breakfast at fasting conditions
  lncRNA expression in count per million measured in blood plasma and whole blood paxgene samples
lncRNA Biomarker expression after breakfast intake | T1- 1 hour after breakfast
  lncRNA expression in count per million measured in blood plasma and whole blood paxgene samples

SECONDARY OUTCOMES:
sncRNA Biomarker expression before breakfast intake | T0- Baseline in the morning before breakfast at fasting conditions
  sncRNA cycle threshold measured in blood plasma
sncRNA Biomarker expression after breakfast intake | T1- 1 hour after breakfast
  sncRNA cycle threshold measured in blood plasma
mRNAs Biomarker expression before breakfast intake | T0- Baseline in the morning before breakfast at fasting conditions
  mRNAs cycle threshold measured in blood plasma
mRNAs Biomarker expression after breakfast intake | T1- 1 hour after breakfast
  mRNAs cycle threshold measured in blood plasma
Soluble proteins Biomarker expression before breakfast intake | T0- Baseline in the morning before breakfast at fasting conditions
  Soluble proteins expression in ng/mL measured in blood plasma
Soluble proteins Biomarker expression after breakfast intake | T1- 1 hour after breakfast
  Soluble proteins expression in ng/mL measured in blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Rohrlich, MD,Phd, Principal Investigator — Firalis SA; Hueseyin Firat, MD, PhD, HDR, Study Director — Firalis SA; Stephanie Boutillier, PhD, Study Chair — Firalis SA
Locations (1):
- Firalis Clinical Investigation Center, Huningue, France

IPD SHARING:
Plan to Share IPD: No